CLINICAL TRIAL: NCT00151489
Title: A Six-Month, Double-Blind, Placebo Controlled, Durability of Effect Study of Pregabalin for Pain Associated With Fibromyalgia
Brief Title: Safety and Efficacy Study of Pregabalin in Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081059
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2006-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin
Drug: placebo

SUMMARY:
The purpose of this research study of pregabalin and fibromyalgia is to see if 1. pregabalin reduces the pain of fibromyalgia and if this effect lasts for six months and 2. to see if different dosages work better (reduce pain and mild to no side effects) for different people.

ELIGIBILITY:
Inclusion Criteria:

* At screening (V1), patients must meet the American College of Rheumatology criteria for fibromyalgia (i.e. widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites
* At Screen (V1) and enrollment (V2), patients must have a score of greater than 40 mm on the Pain Visual Analog Scale

Exclusion Criteria:

* Other severe pain or inflammatory muscle or rheumatologic disease other than fibromyalgia, active infections or untreated endocrine disorders; or severe depression and other serious hepatic, respiratory, hematologic or immunologic illness or active malignancy or history of malignancy (examples of prohibited diseases: Hepatitis C, HIV, diabetes with nerve pain, other nerve pain (shingles), sleep apnea, epilepsy, narcolepsy, rheumatoid arthritis, generalized osteoarthritis, Lupus, Lyme disease unless sign and symptom free for 2 years, Sjogren's Syndrome, Sarcoid, Psoriatic Arthritis, Scleroderma)
* Previous participation in a clinical trial with pregabalin; currently receiving or pending disability claims or workmans compensation or civil litigation, or used other experimental medicines within 30 days of screening
* Creatinine Clearance less than 60 mL/min (estimated from serum creatinine; low platelet and/or white blood cell counts; abnormal Westergren erythrocyte sedimentation rate; abnormal antinuclear antibody (ANA greater than 3U), or rheumatoid factor (RF greater than 80 IU/mL); abnormal (clinically relevant 12 lead ECG)
* Use of prohibited pain/sleep medications (including antidepressants, sedatives, hypnotics, NSAIDs, opiates, muscle relaxants) during the study. Washout required prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020
Dates: Start 2005-04; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of pregabalin (BID) compared with placebo in assessing the durability of effect for the treatment of pain associated with fibromyalgia among patients who initially respond to open-label pregabalin using Pain Visual Analog Scale

SECONDARY OUTCOMES:
To evaluate the efficacy of pregabalin (BID) compared with placebo treatment to relieve pain and to improve global assessment, functional status, sleep and fatigue associated with fibromyalgia using questionnaires. To evaluate the longterm safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (94):
- United States (94):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Calera, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Tuscaloosa, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Stratford, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Palm Springs, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Blue Springs, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Cherry Hill, New Jersey
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, Highland Park, New Jersey
  - Pfizer Investigational Site, Ridgewood, New Jersey
  - Pfizer Investigational Site, South Eddison, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Johnson City, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Smithtown, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Mogadore, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Mechanicsburg, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Sioux Falls, South Dakota
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, South Jordan, Utah
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Charleston, West Virginia

REFERENCES:
- [Derived] Pauer L, Atkinson G, Murphy TK, Petersel D, Zeiher B. Long-term maintenance of response across multiple fibromyalgia symptom domains in a randomized withdrawal study of pregabalin. Clin J Pain. 2012 Sep;28(7):609-14. doi: 10.1097/AJP.0b013e31823dd315. PMID 22688598
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081059&StudyName=Safety+and+Efficacy+Study+of+Pregabalin+in+Fibromyalgia